CLINICAL TRIAL: NCT06140030
Title: Mindfulness-based Stress Reduction in Adolescents With Type 1 Diabetes
Brief Title: Mindfulness Training in Adolescents With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY004827
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Type 1 Diabetes; Quality of Life
MeSH Terms: conditions — Anxiety Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness training mobile health application (Experimental): Use of a mindfulness training mobile health application
  Interventions: Behavioral: Mindfulness training

INTERVENTIONS:
Behavioral: Mindfulness training — Mindfulness-training mobile health application

SUMMARY:
Creation of an adaptation of a mindfulness-based stress reduction mobile health application specifically designed for adolescents living with Type 1 diabetes. Aim to determine whether daily mindfulness improves anxiety symptoms in adolescents with Type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 diabetes for 6 months or longer
* Anxiety score of 5 or higher on the Generalized Anxiety Disorder 7-item scale
* Must be able to read and speak English

Exclusion Criteria:

* Clinical diagnosis of a chronic medical condition requiring intensive daily management

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety Symptoms | 12 weeks
  Generalized Anxiety Disorder 7-item Score range: 0 to 21 Higher scores indicate more anxiety

SECONDARY OUTCOMES:
Diabetes-specific quality of life | 12 weeks
  Pediatric Quality of Life Inventory 3.2 Diabetes Module Range 0 to 100 Higher scores indicate better quality of life
Glycemic control | 12 weeks
  HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida College of Nursing, Tampa, Florida, United States